CLINICAL TRIAL: NCT03043729
Title: mFOLFOX6 vs. mFOLFOX6 + Aflibercept as Neoadjuvant Treatment in MRI-defined T3-rectal Cancer: a Randomized Phase-II-trial
Brief Title: mFOLFOX6 vs. mFOLFOX6 + Aflibercept as Neoadjuvant Treatment in MRI-defined T3-rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Institut für Klinisch-Onkologische Forschung (IKF) Frankfurt (Unknown); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIO-KRK-0214
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Rectal Cancer; Rectosigmoid Cancer
Keywords: neoadjuvant; MRI-defined T3; mFOLFOX6; Aflibercept
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): 6 cycles chemotherapy with Oxaliplatin 85 mg/m^2 and Leucovorin 350 mg/m^2 i.v. as 2h infusion on Day 1 and 5-FU 400 mg/m^2 i.v. as bolus on Day 1 and 2400 mg/m^2 as 46 h infusion q2w followed by surgery 4 weeks after last neoadjuvant chemotherapy treatment
  Interventions: Drug: Oxaliplatin; Drug: 5-FU; Drug: Leucovorin
- Arm B (Experimental): 6 cycles chemotherapy with Oxaliplatin 85 mg/m^2 and Leucovorin 350 mg/m^2 i.v. as 2h infusion on Day 1 and 5-FU 400 mg/m^2 i.v. as bolus on Day 1 and 2400 mg/m^2 as 46 h infusionq2w + Aflibercept 4 mg/kg BW i.v. on Day 1 q2w (6th cycle without Aflibercept) followed by surgery 4 weeks after last neoadjuvant chemotherapy treatment
  Interventions: Drug: Oxaliplatin; Drug: 5-FU; Drug: Leucovorin; Biological: Aflibercept

INTERVENTIONS:
Drug: Oxaliplatin — Oxaliplatin 85 mg/m^2, as 2h infusion on Day 1 (Arm A + Arm B)
Drug: 5-FU — 5-FU 400 mg/m^2 i.v. as bolus on Day 1 and 2400 mg/m^2 as 46 h infusion q2w (Arm A + Arm B)
Drug: Leucovorin — Leucovorin 350 mg/m^2 i.v. as 2h infusion on Day 1 (Arm A + Arm B)
Biological: Aflibercept — Aflibercept 4 mg/kg BW i.v. on Day 1 q2w (Arm B, Cycles 1 to 5)
  Arms: Arm B

SUMMARY:
Patients with locally advanced rectal or rectosigmoid cancer staged cT3 CRM-negative with MRI will receive 6 cycles of neoadjuvant treatment with mFOLFOX6 (Arm A) vs. mFOLFOX6 + aflibercept (Arm B) followed by surgery.

DETAILED DESCRIPTION:
Patients with locally advanced rectal cancer are generally recommended to receive preoperative radiotherapy or radiochemotherapy. The advantage of combined-modality therapy in rectal cancer is that it has reduced local pelvic recurrence - a dreaded and morbid event - to rates of about 10%. There is good quality evidence that preoperative radiotherapy reduces local recurrence but there is little if any impact on overall survival. One strategy to reduce the distant recurrence rate, and thereby increase the cure rate, would be to introduce systemic treatment earlier to prevent dissemination of micrometastases. The present trial is designed to compare two neoadjuvant chemotherapy regimens in patients with non-metastatic T3 CRM-negative rectal cancers using quality-controlled MRI of the pelvis as a main inclusion criterion. This strategy is believed to reduce acute and long-term toxicity caused by preoperative radiotherapy and to administer effective systemic chemotherapy early in the course of disease as neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years on day of signing informed consent
2. Signed and dated informed consent, and willing and able to comply with protocol requirements
3. WHO/ECOG Performance Status (PS) 0-1
4. Diagnosis of rectal adenocarcinoma
5. Candidate for sphincter-sparing surgical resection prior to neoadjuvant therapy according to the primary surgeon, i.e. no patient will be included for whom surgeon indicates need for abdomino-perineal resection (APR) at baseline.
6. Clinical staging is based on the combination of the following assessments:

   * Physical examination by the primary surgeon
   * CT scan of the chest/abdomen
   * Pelvic MRI
   * Rigid rectoscopy / endoscopic ultrasound (ERUS).
   * Both examinations (i.e. MRI and ERUS) are mandatory.
7. The tumor has to fulfill the following criteria:

   * No symptomatic bowel obstruction
   * Locally advanced rectal and rectosigmoid cancer, i.e. lower border of tumor > 5 cm and < 16 cm from anal verge as determined by rigid rectoscopy
   * MRI criteria:

     1. Lower border of tumor below a line defined by promontorium and symphysis, regardless of the criterion "< 16 cm from anal verge as determined by rigid rectoscopy".
     2. No evidence that tumor is adjacent to (defined as within 2 mm of) the mesorectal fascia on MRI (i.e. CRM > 2 mm)
     3. Only T3-tumors are included, i.e infiltration into perirectal fat < 10 mm provided CRM > 2 mm
     4. Note: MRI criteria are used for the definition of T3 tumor (i.e. exclusion of T2 and T4 situation).
8. Hematological status:

   * Neutrophils (ANC) ≥ 2 x 10^9/L
   * Platelets ≥ 100 x 10^9/L
   * Hemoglobin ≥ 9 g/dL (previous transfusion of packed blood cells allowed)
9. Adequate renal function:

   * Serum creatinine level ≤ 1.5 x upper limit normal (ULN) or ≤ 1.5 mg/dl
   * Creatinine clearance ≥ 30 ml/min
10. Adequate liver function:

    * Serum bilirubin ≤ 1.5 x upper limit normal (ULN)
    * Alkaline phosphatase < 3 x ULN
    * AST and ALT < 3 x ULN
11. Proteinuria < 2+ (dipstick urinalysis) or ≤ 1 g/24hour or ≤ 500mg/dl
12. Regular follow-up feasible
13. For female patients of childbearing potential, negative pregnancy test within 1 week (7 Days) prior of starting study treatment
14. Female patients of childbearing potential (i.e. did not undergo surgical sterilization - hysterectomy, bilateral tubal ligation, or bilateral oophorectomy - and is not post-menopausal for at least 24 consecutive months) must commit to using high effective and appropriate methods of contraception until at least 6 months after the end of study treatment such as combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomized partner, sexual abstinence. If an oral contraception is used, a barrier method of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge) has to be applied additionally
15. Fertile male patients with a partner of childbearing potential must commit to using high effective and appropriate methods of contraception (details see above) until at least 9 months after the end of study treatment.

Exclusion Criteria:

1. Distant metastases (CT scans of thorax and abdomen are mandatory)
2. cT2 and cT4 tumors (defined by MRI criteria)
3. Exclusion of potentially compromised CRM as defined by MRI criteria (i.e. > 2 mm distance from CRM)
4. Prior antineoplastic therapy for rectal cancer
5. History or evidence upon physical examination of CNS metastasis
6. Uncontrolled hypercalcemia
7. Pre-existing permanent neuropathy (NCI-CTCAE grade ≥ 2)
8. Uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy
9. Concomitant protocol unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy, radiotherapy)
10. Treatment with any other investigational medicinal product within 28 days prior to study entry
11. Known dihydropyrimidine dehydrogenase (DPD) deficiency
12. Treatment with CYP3A4 inducers unless discontinued > 7 Days prior to randomization
13. Any of the following in 3 months prior to inclusion:

    * Grade 3-4 gastrointestinal bleeding
    * Treatment resistant peptic ulcer disease
    * Erosive esophagitis or gastritis
    * Infectious or inflammatory bowel disease
    * Diverticulitis
14. Any active infection within 2 weeks prior to study inclusion
15. Vaccination with a live, attenuated vaccine within 4 weeks prior to the first administration of the study medication
16. Other concomitant or previous malignancy, except:

    * Adequately treated in-situ carcinoma of the uterine cervix
    * Basal or squamous cell carcinoma of the skin
    * Cancer in complete remission for > 5 years
17. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days prior to study entry
18. Pregnant or breastfeeding women
19. Patients with known allergy to any constituent to study drugs
20. History of myocardial infarction and/or stroke within 6 months prior to randomization, NYHA class III and IV congestive heart failure
21. Severe renal insufficiency (creatinin clearance < 30 ml/min)
22. Bowel obstruction
23. Contra-indication to the assessment by MRI
24. Involvement in the planning and/or conduct of the study (applies to both Sanofi staff and/or staff of Sponsor and study site)
25. Patient who might be dependent on the sponsor, site or the investigator
26. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 AMG
27. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | 20 weeks
  number of patients with a pCR finding divided by the number of patients in the analysis set pCR will be assessed in a standardized manner independently by a central pathology

SECONDARY OUTCOMES:
Dose intensities of study medication | 12 weeks
  The dose intensities of study medication will be calculated over the whole study duration and will be summarized descriptively by summary statistics.
Type, incidence and severity of AEs, SAEs | 20 weeks
  AEs will be coded according to the NCI-CTC Criteria Version 4.03. For the analysis, all AEs will be classified as related and not related. AEs will be summarized by presenting the number and percentages of patients having any AE and having an AE in each NCI-CTC category. Summaries will also be presented for AEs by severity and relationship to study medication. Tables will be broken down by study arm. All deaths and serious adverse events will be listed and briefly described.
Dose reduction or discontinuation of study drug due to adverse events | 20 weeks
  The dose intensities of study medication will be calculated over the whole study duration and will be summarized descriptively by summary statistics.
Rate of treatment discontinuation due to toxicity | 20 weeks
  Summaries will also be presented for AEs by severity and relationship to study medication. Tables will be broken down by study arm.
  All deaths and serious adverse events will be listed and briefly described.
Type, incidence and severity of laboratory abnormalities | 20 weeks
  For relevant laboratory parameters, the distribution over time as well as changes from randomization will be calculated and analyzed descriptively.
Rate of patients with R0-wide resection (according to CRM definitions in S3 guideline-Version 1.1 August 2014) | 20 weeks
  The R0- and R1 resection as well as downstaging and downsizing using a standardized regression grading (Dworak regression grading) will be analyzed descriptively by means of frequencies and percentages.
Rate of patients with R0-narrow resection (according to CRM definitions in S3 guideline-Version 1.1 August 2014) | 20 weeks
  The R0- and R1 resection as well as downstaging and downsizing using a standardized regression grading (Dworak regression grading) will be analyzed descriptively by means of frequencies and percentages.
Rate of patients with R1 resection (according to CRM definitions in S3 guideline-Version 1.1 August 2014) | 20 weeks
  The R0- and R1 resection as well as downstaging and downsizing using a standardized regression grading (Dworak regression grading) will be analyzed descriptively by means of frequencies and percentages.
Rate of patients with locoregional R2 resection (according to CRM definitions in S3 guideline-Version 1.1 August 2014) | 20 weeks
  The R0- and R1 resection as well as downstaging and downsizing using a standardized regression grading (Dworak regression grading) will be analyzed descriptively by means of frequencies and percentages.
Rate of number of patients with R0-wide, R0-narrow (according to CRM definitions in S3 guideline-Version 1.1 August 2014), R1 and locoregional R2 resection | 20 weeks
  The R0- and R1 resection as well as downstaging and downsizing using a standardized regression grading (Dworak regression grading) will be analyzed descriptively by means of frequencies and percentages.
Disease-free survival (DFS) | 44 weeks
  Disease-free survival rate will be analyzed using a two-sided Fisher's exact test at a 5% significance level. In addition, two-sided 95% confidence intervals for DFS rates and difference in rates between both treatment arms will be calculated.
Relapse-free survival (RFS) in resected patients | 44 weeks
  Relapse-free survival: The length of time after completion of primary treatment (neoadjuvant chemotherapy + surgery) until documented relapse (i.e. local relapse, liver metastasis, systemic metastases).
Overall survival (OS) rate | 44 weeks
  Overall survival: Survival will be calculated from the date of subject enrollment until the date of death from any cause. If no event is observed (e.g. lost to follow-up) OS is censored at the day of last subject contact.
Downstaging ability in resected patients using a standardized regression grading (Dworak regression grading) | 20 weeks
  The R0- and R1 resection as well as downstaging and downsizing using a standardized regression grading (Dworak regression grading) will be analyzed descriptively by means of frequencies and percentages.
Downsizing ability in resected patients using a standardized regression grading (Dworak regression grading) | 20 weeks
  The R0- and R1 resection as well as downstaging and downsizing using a standardized regression grading (Dworak regression grading) will be analyzed descriptively by means of frequencies and percentages.
Type, incidence and severity of perioperative medical events within 28 days after surgery are assessed. Perioperative morbidity is categorized according to the Clavien-Dindo-Classification | 20 weeks
  Perioperative medical events as well as mortality within 28 days after surgery will be summarized by frequencies and percentages broken down per treatment arm.
Mortality after surgery | 20 weeks
  Perioperative medical events as well as mortality within 28 days after surgery will be summarized by frequencies and percentages broken down per treatment arm.
Vital signs | 20 weeks
  Vital signs will be analyzed using summary statistics broken down per treatment group and visit.
Physical examination | 20 weeks
  Physical examination as well as WHO/ECOG will be analyzed by calculating frequencies and percentages broken down per treatment group and visit.
ECOG | 20 weeks
  Physical examination as well as WHO/ECOG will be analyzed by calculating frequencies and percentages broken down per treatment group and visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf-Dieter Hofheinz, Prof. Dr., Principal Investigator — Tagestherapiezentrum am ITM & III. Med. Klinik, Universitätsmedizin Mannheim
Locations (1):
- Tagestherapiezentrum am ITM & III. Med. Klinik, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No